CLINICAL TRIAL: NCT04448184
Title: Platelet Transfusions in Hematopoietic Stem Cell Transplantation - The PATH Phase III Trial
Brief Title: Platelet Transfusions in Hematopoietic Stem Cell Transplantation (The PATH III Trial)
Acronym: PATH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Alberta Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2068
Record Dates: First submitted 2020-04-24; First posted 2020-06-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic Platelet Transfusion (No Intervention): Patients allocated to the prophylactic platelet transfusion group will receive a platelet transfusion when the measured platelet count is less than 10 x 109/L.
- Prophylactic Tranexamic Acid (Experimental): Patients allocated to the prophylactic Tranexamic Acid group will receive a standardized routine oral or intravenous dose of Tranexamic Acid 1 gram three times daily.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Patients allocated to the prophylactic Tranexamic Acid group will receive a standardized routine oral or intravenous dose of Tranexamic Acid 1 gram three times daily.
  Tranexamic Acid will start when Platelet count is less than 50 x 109/L and continue until platelet engraftment. Patients in this group will not receive routine prophylactic platelet transfusions. Subjects unable to swallow oral Tranexamic Acid pills may have the tablets crushed, administered via nasogastric (NG) tube or the medication will be administered intravenously.
  Other Names: SteriMax Inc.; Cyclokapron®
  Arms: Prophylactic Tranexamic Acid

SUMMARY:
It is hypothesized that a strategy using prophylactic oral and intravenous Tranexamic Acid (TXA) with therapeutic platelet transfusions (if required) is safe and more effective than prophylactic platelet transfusions in patients undergoing an autologous hematopoietic stem cell transplantation (ASCT).

DETAILED DESCRIPTION:
In Canada, over 1,500 autologous hematopoietic stem cell transplantations (ASCT) are performed annually for hematologic malignancies. It is currently standard practice to provide a prophylactic transfusion of platelets to prevent bleeding when the daily measured platelet count is less than 10 x 109/L. A patient may require up to six adult platelet doses during the post-transplant period. However, the true benefit of prophylactic platelet transfusions in the ASCT setting is unclear and has been called into question by several recent studies.

Prophylactic platelet transfusions may not only be unnecessary, they may be detrimental to the patient. Among blood products, platelet transfusions are associated with the highest risk of both infectious and non-infectious complications: this would include bacterial infections and allergic /febrile reactions. Moreover, the potential overuse of platelet products places a significant burden on a scarce health care resource that is provided through volunteer donations.

An alternative strategy to prevent bleeding and reduce the need for platelet transfusions involves administering Tranexamic Acid, an antifibrinolytic agent to stabilize blood clots and reduce bleeding. Tranexamic Acid is safe and effective in many clinical scenarios, and may be a reasonable alternative for prophylactic platelet transfusions. In the setting of ASCT, Tranexamic Acid may reduce bleeding and further enhance a strategy of therapeutic platelet transfusions where platelets are administered only in the event of active bleeding symptoms.

The effect of prophylactic platelet transfusions and Tranexamic Acid on clinical, quality of life and economic outcomes in patients receiving ASCT is unknown. The primary aim of this research program is to perform a randomized controlled trial to determine whether a strategy of prophylactic Tranexamic Acid (with therapeutic platelet transfusions) is safe and effective compared to prophylactic platelet transfusions in patients undergoing ASCT.

A pilot trial demonstrated feasibility by successfully recruiting 100 patients and these patients will be rolled over into the phase III study. The treatment assignment and bleeding outcomes for these patients remain blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years or older undergoing ASCT for a hematologic malignancy
2. Patients providing written informed consent prior to starting transplantation

Exclusion Criteria:

1. A previous WHO grade 2, 3 or 4 bleeding event within the past year
2. A previous or current unprovoked thrombotic event defined as a pulmonary embolism, deep vein thrombosis, cerebral thrombosis
3. A current provoked thrombotic event (e.g. catheter-related thrombosis) within last month and/or still requiring anticoagulant treatment.
4. A requirement for therapeutic anticoagulant or anti-platelet drugs during ASCT
5. Active angina (chest pain of presumed cardiac origin either at rest or with activity)
6. Current or previous (within 2 weeks) urinary tract bleeding
7. An inherited hemostatic or thrombotic disorder
8. Coagulopathy defined as a prothrombin time '/International Normalization Ratio (INR) or activated partial thromboplastin time more than 1.5 times the upper limit of normal or fibrinogen less than 2 g/L
9. Previously documented history of refractoriness to platelet transfusion secondary to HLA antibodies (Refractoriness is defined as 2 consecutive ABO matched platelet transfusions with platelet increment of < 7.5 and the presence of anti-HLA antibodies)
10. Significant renal impairment (creatinine more than 1.5 times the upper limit of normal or a eGFR less than 0.5 mL/min/1.78m2)
11. Pregnant or breast-feeding
12. Unwilling or unable to provide informed consent
13. Participant has acquired disturbances to his/her colour vision (does not apply to congenital colour blindness)
14. Participant has known sensitivity or allergy to Tranexamic Acid or any of its ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 662 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
WHO (World Health Organization) bleeding events of Grade 2 or higher | Daily, up to 30 days

SECONDARY OUTCOMES:
WHO bleeding events of Grade 3 or 4 | Daily, up to 30 days
Time from randomization to bleeding of WHO events Grade 2 or higher | Daily, up to 30 days
Number of days with bleeding of WHO bleeding events Grade 2 or higher | Daily, up to 30 days
Bleeding Severity Measurement Scale (BSMS) for bleeding events Grade 2 or higher | Daily, up to 30 days
  The BSMS scale measures bleeding grade and classification from 0-2. 0 indicates no bleeding. Grade 1 bleeding consists of trace bleeding and mild bleeding and is not clinically significant. Grade 2 bleeding consists of serious bleeding, serious bleeding causing significant morbidity, and fatal bleeding. Grade 2 bleeding is clinically significant.
Number of platelet and/or red blood cell transfusions | Daily, up to 30 days
Adverse reactions related to tranexamic acid | Daily, up to 30 days.
  Number and type of reactions will be recorded.
Venous thromboembolism grade 2 or higher | Daily, up to 30 days.
Adverse reactions related to platelet transfusion | Daily, up to 30 days.
  Number and type of reactions will be recorded.
Time to platelet count recovery | Daily, up to 30 days.
Number of days with a platelet count < 10 x 109/L | Daily, up to 30 days.
LOS (Length of hospital stay) | LOS will be measured as the number of days elapsed between hospital admission and hospital discharge date up to 30 days.
  LOS = admission date - discharge date
Transplant related outcome: Bearman Scoring System for Organ Toxicity following HSCT | Day 30
  This is a validated scoring system to assess toxicity during HSCT. In this system, grade I toxicity is reversible without treatment and grade 2 is not life threatening, but requires treatment. Grade 3 requires life-support intervention and grade 4 is fatal. Regimen-related toxicity in each organ system was scored as the highest grade achieved in that organ system through day 28, except that deaths occurring after day 28 as a result of regimen-related toxicity occurring before day 28 are also scored as grade 4. Adverse events that could be attributed to infection (culture-documented), bleeding or other medications are not scored as regimen-related toxicity. The maximum toxicity is the highest grade recorded in any individual organ system and the cumulative toxicity score is the sum of the highest grades recorded for all eight organ systems.
Transplant related outcome: Incidence of infections at Day 30 following ASCT | Day 30
Transplant related outcome: Mortality at Day 30 and 180 | Day 30, Day 180
Economic Analyses | 5 years
  Incremental cost effectiveness ratios
Quality of Life Measure: FACT-Thrombocytopenia 18 | Weekly, up to 30 days
  The FACT consists of 5 subscales that measure physical well-being, functional well-being, social/family well-being and emotional well-being. The BMT subscale of the FACT includes additional items specifically designed to test quality of life and symptoms specific to transplant patients.
Quality of Life Measure: FACT- BMT | Day 30, Day 90, Day 180
  The FACT-BMT scale is valid and sensitive to clinical change in transplant recipients. It is the most consistently used scale amongst the Canadian Bone Marrow Transplant Group (CBMTG). It is the preferred scale in several Canadian multicentre trials in stem cell transplantation. FACT- Thrombocytopenia 18 is valid measure to elicit quality of life due to thrombocytopenia, and will complement the FACT-BMT scale.
Quality of Life Measure: GAD-7 | Weekly, up to 30 days
  GAD-7 is a short validated scale that assesses symptoms of generalized anxiety and is commonly used in medical settings. There is no specific validated scale to assess anxiety of patients who are at risk for bleeding.
Quality of Life Measure: EQ-5D | Weekly, up to 30 days
  EQ-5D is a standardized measure of health status to provide a simple, generic measure of health for clinical and economic appraisal. It is applicable to a wide range of health conditions and treatments; it provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health care. It is cognitively undemanding, taking only a few minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Tinmouth, MD, Principal Investigator — The Ottawa Hospital
Locations (12):
- Canada (12):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Eastern Regional Health Authority, St. John's, Newfoundland and Labrador
  - Memorial University, St. John's, Newfoundland and Labrador
  - Dalhousie University, Halifax, Nova Scotia
  - Hamilton Health Sciences - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Saskatchewan Cancer Agency, Saskatoon, Saskatchewan